CLINICAL TRIAL: NCT07028918
Title: Phase II Trial of Neoadjuvant Chemoimmunotherapy With Low-Dose Radiotherapy in Locally Advanced Oral Squamous Cell Carcinoma: A Prospective Single-Arm Study
Brief Title: A Prospective Single-Arm Study（NCLDR）
Acronym: NCLDR
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202502-008-1
Record Dates: First submitted 2025-06-01; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Oral Squamous Cell Carcinoma (OSCC)
Keywords: Phase III, IVA, and IVB
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Acidemia, isovaleric | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OSCC（III、IVA、IVB） (Experimental): Patients with locally advanced oral squamous cell carcinoma (clinical stages III, IVA, and IVB according to AJCC clinical staging)
  Interventions: Radiation: Low dose radiotherapy regimen; Drug: New adjuvant immunotherapy regimen; Procedure: Surgical treatment; Drug: Postoperative adjuvant therapy plan; Radiation: Radical radiotherapy plan

INTERVENTIONS:
Radiation: Low dose radiotherapy regimen — On the first and second day of chemotherapy and immunotherapy, low-dose radiotherapy of 1 Gy/1f was administered to the primary tumor lesion and metastatic lymph nodes, respectively, for a total of 4 Gy/4f.
Drug: New adjuvant immunotherapy regimen — Terriptylimab: fixed dose 240 mg, q30000, intravenous infusion, each infusion lasting 30 minutes (not less than 20 minutes, not more than 60 minutes); Chemotherapy regimen: Albumin bound paclitaxel: 175-260 mg/m2, d1, q3w; Platinum class: Cisplatin: 75mg/m2, d1-3, q3w; Carboplatin: AUC=5, d1, q3w (for patients with cisplatin allergy, intolerance, hearing impairment, creatinine clearance rate<50ml/min, or grade 1 neuropathy that are not suitable for cisplatin use).
Procedure: Surgical treatment — Surgery begins around 4 weeks after the first day of the second cycle of neoadjuvant therapy. The surgical plan is developed and evaluated by oral surgeons with years of clinical surgical experience. The determination of surgical margins is mainly based on baseline standards before neoadjuvant therapy for tumors, and can be appropriately reduced by oral surgeons depending on the situation.
Drug: Postoperative adjuvant therapy plan — * Patients with postoperative pathological progression of pCR were given maintenance treatment with Triprolizumab Q3W for 1 year.
    * Patients with postoperative pathology not reaching pCR should receive adjuvant radiotherapy (60-66Gy/30-33f) ③ Patients with high-risk recurrence factors in postoperative pathology (positive tumor margin or insufficient safe margin, presence of lymph node extracellular invasion) are given adjuvant radiotherapy and chemotherapy.
Radiation: Radical radiotherapy plan — ① Radical radiotherapy for the primary lesion and cervical lymphatic drainage area.
  ② Synchronous cisplatin during radiotherapy: 75mg/m2, d1-3, q3w.

SUMMARY:
To investigate the safety and efficacy of low-dose radiotherapy combined with chemotherapy and immunotherapy as neoadjuvant therapy for locally advanced oral squamous cell carcinoma (OSCC), and to explore whether low-dose radiotherapy can induce cross-presentation of tumor-specific antigens, enhance lymphocyte infiltration into the tumor microenvironment, and thereby amplify tumor-specific immune responses, ultimately improving the therapeutic outcomes of neoadjuvant chemoimmunotherapy.

DETAILED DESCRIPTION:
This study is a prospective, phase II clinical trial that enrolled patients with locally advanced oral squamous cell carcinoma (based on AJCC clinical staging, clinical stages III, IVA, and IVB). The patients were treated with a combination of albumin paclitaxel and cisplatin and trastuzumab for 2 cycles before surgery. On the day of the 2 chemotherapy immunotherapy sessions and the second day (d1, d2), the patients were given 1 Gy/1f of radiation therapy for the primary lesion and metastatic lymph nodes, for a total of 4 Gy/4f. Approximately 4 weeks after the first day of the second treatment cycle, evaluate the condition of the lesion and cervical lymph nodes. Patients can undergo surgical treatment after resection. After surgery, based on pathological results, decide on the postoperative adjuvant treatment plan: patients with postoperative pathological progression of pCR will receive maintenance treatment with Triprolizumab Q3W for 1 year, while patients without postoperative pathological progression of pCR will receive adjuvant radiotherapy (60-66Gy/30-33f). If there are high-risk recurrence factors (positive tumor margin or insufficient safe margin, lymph node extracellular invasion), adjuvant radiotherapy and chemotherapy will be given. Patients assessed as unresectable will receive curative radiotherapy and chemotherapy, and immune maintenance will be chosen based on the patient's specific condition after completion. Collect safety related indicators such as adverse reactions (AE) and surgical delay rate during and after treatment for patients; pCR、MPR、 Use treatment related indicators such as 2-year EFS rate, 2-year OS rate, and oral function retention rate to statistically analyze the effectiveness and safety of treatment plans.

ELIGIBILITY:
【Inclusion Criteria】:

1. Age: 18 to 70 years old (inclusive) at the time of enrollment, based on the Gregorian calendar birth date. Age calculation is based on the date of signing the informed consent form. Includes both males and females.
2. ECOG Performance Status: 0-1.
3. Life Expectancy: ≥ 6 months.
4. Diagnosis: Histologically confirmed oral squamous cell carcinoma.
5. Clinical Stage: Stage III, IVA, or IVB according to AJCC clinical staging.
6. Absence of Distant Metastasis: No evidence of distant metastasis confirmed by auxiliary examinations.
7. Prior Anti-tumor Therapy: No previous surgery, radiotherapy, chemotherapy, immunotherapy, targeted therapy, or other anti-tumor treatments.
8. Measurable Lesion: At least one measurable target lesion according to RECIST 1.1 criteria, confirmed by imaging during the screening period.
9. Adequate Organ Function: Meeting the following criteria:

   * Hematology: White blood cell count (WBC) ≥ 4.0 x 10⁹/L; Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L; Hemoglobin (Hb) ≥ 90 g/L; Platelets (PLT) ≥ 100 x 10⁹/L.
   * Liver Function: ALT and AST < 3 x Upper Limit of Normal (ULN); Total bilirubin < 1.5 x ULN; Child-Pugh class A or B; Normal liver tissue volume ≥ 700 cm³.
   * Renal Function: Serum creatinine < 1.5 x ULN.
   * Coagulation: International Normalized Ratio (INR) and Activated Partial ·Thromboplastin Time (APTT) ≤ 1.5 x ULN.
   * Serum Albumin: ≥ 28 g/L.
   * Urinalysis: Urine protein < 2+ (If baseline urine protein ≥ 2+, a 24-hour urine protein quantification must be performed within 7 days; enrollment requires quantification < 1g).
   * Electrocardiogram (ECG): No significant abnormalities.
   * Cardiac Function: Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
10. Contraception: Women of childbearing potential must have reliable contraception or have a negative pregnancy test (serum or urine) within 7 days prior to enrollment. They must be willing to use adequate contraception during the trial and for 8 weeks after the last dose of the study drug. Men must agree to use adequate contraception or be surgically sterilized during the trial and for 8 weeks after the last dose of the study drug.
11. Informed Consent: Ability to understand and voluntarily sign the informed consent form (signed by a legal representative if the participant loses capacity), with expected good compliance.

【Exclusion Criteria】:

1. Unsuitable for Treatment: Unsuitable for receiving the protocol-specified low-dose radiotherapy, immunotherapy, and chemotherapy.
2. Prior Anti-tumor Therapy: Previous treatment with anti-tumor therapy, including investigational drugs, chemotherapy, radiotherapy, or prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2 antibodies/drugs, or any other antibody/drug specifically targeting T-cell co-stimulatory checkpoint pathways.
3. Active Infection: Severe active infection requiring systemic therapy.
4. Cardiovascular/Cerebrovascular Events: History within 6 months prior to study treatment of: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism.
5. Bleeding Tendency/Disorder: Definite bleeding tendency or clinically significant bleeding symptoms within 28 days, including but not limited to gastrointestinal bleeding, epistaxis (excluding minor nosebleeds and blood-tinged sputum), or ongoing hemorrhagic or coagulopathic disease.
6. Systemic Corticosteroids: Requirement for systemic corticosteroid therapy (>10 mg/day prednisone or equivalent dose) or replacement therapy (>10 mg/day prednisone equivalent) within 14 days prior to study treatment.
7. Recent Procedures: Live vaccination within 4 weeks prior to study treatment or planned during the study period. Major surgery within 4 weeks prior to study treatment.
8. Pregnancy/Lactation: Pregnant or breastfeeding women.
9. Infectious Disease:

   * Known immunodeficiency.
   * Known history of Human Immunodeficiency Virus (HIV) or Acquired --·Immunodeficiency Syndrome (AIDS)-defining illness.
   * Hepatitis B Virus (HBV) infection (HBsAg positive) or Hepatitis C Virus (HCV) ·infection (HCV RNA positive if anti-HCV antibody screening is positive).
   * Known active history of Tuberculosis (TB).
10. Other Exclusionary Conditions: Any other factor identified by the investigator that may lead to premature termination of the study, such as severe laboratory abnormalities, or concomitant familial or social factors that could compromise participant safety or affect data/sample collection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Complete pathological response rate | Surgery completed based on pathological results，9-10 week
  Complete pathological response rate (pCR) of low-dose radiotherapy combined with chemotherapy and immune neoadjuvant therapy for locally advanced oral squamous cell carcinoma patients

SECONDARY OUTCOMES:
Failure to achieve pathological remission rate (pCR) | 2 year
  Secondary endpoints: The major pathological response (MPR) rate, objective response rate (ORR), oral function preservation rate, 2-year event-free survival (EFS) rate, 2-year overall survival (OS) rate, and safety profile of low-dose radiotherapy combine

IPD SHARING:
Plan to Share IPD: No
1. Ethical restrictions prohibiting open data sharing per local IRB.
  2. Inclusion of potentially identifiable biometric data.